CLINICAL TRIAL: NCT06492577
Title: Effectiveness of Combined Pulmonary Rehabilitation and Progressive Muscle Relaxation on Long-term COVID-19 Symptoms: a Randomized Controlled Trial
Brief Title: Combined Pulmonary Rehabilitation and PMR for Long-Term COVID-19 Symptoms: A RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spitalul Clinic de Boli Infecțioase și Pneumoftiziologie Dr. Victor Babeș Timișoara (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4990
Record Dates: First submitted 2024-07-04; First posted 2024-07-09 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Long Covid19; Pulmonary Rehabilitation; Progressive Muscle Relaxation
Keywords: Long-COVID-19; Progressive Muscle Relaxation; Pulmonary Rehabilitation; Exercise Capacity; Anxiety Reduction
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary rehabilitation group (Active Comparator): Participants in this arm will undergo a structured 21-day pulmonary rehabilitation (PR) program designed to improve lung function, exercise capacity, and overall physical health, conducted according to the American Thoracic Society (ATS) guidelines. The program includes aerobic exercises performed five days per week at moderate intensity (4-6 on the Borg RPE scale) for 30-45 minutes per session, including warm-up and cool-down periods. Strength training will be conducted three days per week on non-consecutive days, starting at 50% of the one-repetition maximum (1RM) and progressively increasing to 70% as tolerated, with each session lasting 20-30 minutes and including 2-3 sets of 8-12 repetitions for major muscle groups. Daily breathing exercises focusing on controlled techniques such as diaphragmatic and pursed-lip breathing will be performed for 10-15 minutes per session.
  Interventions: Other: Pulmonary rehabilitation protocol
- Progressive muscle relaxation group (Experimental): Participants in this group will receive additional progressive muscle relaxation techniques designed to reduce anxiety and improve sleep quality in patients with long-term COVID-19 symptoms. Each PMR session will last for 20 minutes and will involve systematic muscle tensing and relaxation, starting from the feet and progressing to the head, combined with slow, deep breathing.
  Interventions: Other: Pulmonary rehabilitation protocol; Other: Progressive muscle relaxation protocol

INTERVENTIONS:
Other: Pulmonary rehabilitation protocol — In the initial phase (days 1-7), aerobic exercise sessions will be 20-30 minutes, strength training will include 1-2 sets at 50% of 1RM, and breathing exercises will last 10 minutes daily. In the progressive phase (days 8-14), aerobic exercise sessions will increase to 30-40 minutes, strength training to 2-3 sets at 60% of 1RM, and breathing exercises to 10-15 minutes daily. In the advanced phase (days 15-21), aerobic exercise sessions will be 40-45 minutes, strength training will be 2-3 sets at 70% of 1RM, and breathing exercises will continue for 10-15 minutes daily.
Other: Progressive muscle relaxation protocol — Participants in this arm will undergo a 21-day progressive muscle relaxation (PMR) program aimed at reducing anxiety and improving sleep quality in patients with long-term COVID-19 symptoms. Each daily session lasts 20 minutes and involves systematic muscle tensing and relaxation, starting from the feet and progressing to the head, combined with slow, deep breathing. During the initial phase (days 1-7), the focus is on introducing PMR techniques and targeting different muscle groups. In the progressive phase (days 8-14), full-body PMR sessions enhance relaxation and breathing techniques. The advanced phase (days 15-21) maximizes relaxation and incorporates visualization techniques.
  Arms: Progressive muscle relaxation group

SUMMARY:
Our study aimed to evaluate the effectiveness of a 21-day program combining pulmonary rehabilitation (PR) with progressive muscle relaxation (PMR) in patients experiencing long-term symptoms of COVID-19. Participants with persistent symptoms will be randomly assigned to either a PR group or a PR combined with PMR group. The PR program includes aerobic exercises, strength training, and breathing exercises, while the PMR sessions involve systematic muscle tensing and relaxation techniques. We will measure outcomes such as lung function, exercise capacity, anxiety, depression, and sleep quality using validated questionnaires and clinical tests.

DETAILED DESCRIPTION:
The study aims to evaluate the effectiveness of a 21-day combined pulmonary rehabilitation (PR) and progressive muscle relaxation (PMR) program on improving physical and psychological outcomes in patients with long-term COVID-19 symptoms.

This is a parallel, randomized controlled trial (RCT) with two intervention groups: a pulmonary rehabilitation (PR) group and a PR combined with progressive muscle relaxation (PR + PMR) group.

The study will enroll adults aged 18-75 with persistent moderate to severe long-term COVID-19 symptoms, specifically dyspnea and fatigue, lasting at least three months post-infection. Inclusion criteria include confirmed COVID-19 diagnosis via PCR or antibody tests, stable medical condition, and mental readiness to participate. Exclusion criteria include severe comorbid conditions, recent major surgery, severe cognitive or psychiatric disorders, active respiratory infections, severe mobility impairments, and high alcohol or substance abuse.

Participants in the PR group will undergo a 21-day pulmonary rehabilitation program designed to improve lung function, exercise capacity, and overall physical health, following American Thoracic Society (ATS) guidelines. The program includes aerobic exercises performed five days per week at moderate intensity (4-6 on the Borg RPE scale) for 30-45 minutes per session, including warm-up and cool-down periods. Strength training is conducted three days per week on non-consecutive days, starting at 50% of the one-repetition maximum (1RM) and progressively increasing to 70% as tolerated, with each session lasting 20-30 minutes and including 2-3 sets of 8-12 repetitions for major muscle groups. Daily breathing exercises focusing on controlled techniques such as diaphragmatic and pursed-lip breathing for 10-15 minutes per session.

In addition to the PR program, participants in the PR + PMR group will perform daily PMR sessions designed to reduce anxiety and improve sleep quality. Each PMR session will last 20 minutes, involving systematic muscle tensing and relaxation starting from the feet and progressing to the head, combined with slow, deep breathing.

The primary outcomes include lung function, exercise capacity, anxiety, depression, sleep quality, and psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COVID-19 through documented positive PCR or antibody tests.
* Persistent long-COVID-19 symptoms, specifically moderate or severe dyspnea and fatigue, lasting for at least three months post-infection.
* Adults aged between 18 and 75 years.
* Stable medical condition with no recent exacerbations or hospital admissions for other conditions in the past three months.

Exclusion Criteria:

* Severe comorbid conditions such as moderate to severe heart disease, severe ischemic or hemorrhagic stroke, neurodegenerative diseases, or severe acute illnesses.
* Major surgery or hospitalization for severe conditions within the past six months.
* Severe cognitive or psychiatric disorders, determined through comprehensive cognitive and psychiatric evaluations.
* Active respiratory infections or immunocompromised status.
* Severe mobility impairments or chronic pain that could limit participation in rehabilitation exercises.
* High alcohol intake or substance abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Lung function | 20 minutes
  Spirometry is a pulmonary function test used to assess lung function by measuring the volume and speed of air that can be inhaled and exhaled. During the procedure, the patient sits upright, uses a nose clip, and takes a deep breath in. They then exhale as forcefully and quickly as possible into a spirometer through a disposable mouthpiece. This process measures the maximum volume of air expelled (Forced Vital Capacity, FVC) and the volume expelled in the first second (Forced Expiratory Volume in One Second, FEV1). The test is repeated at least three times to ensure accuracy, and the best effort is recorded.
Exercise capacity | 20 minutes
  The exercise capacity evaluation will be conducted using the 6-minute walk test (6MWT). During the test, the patient is instructed to walk back and forth along a flat, straight 30-meter course for six minutes, aiming to cover as much distance as possible. The total distance walked in six minutes is measured in meters. Rest periods are allowed if necessary, but the clock continues to run.
Anxiety | At inclusion and at the end of the study
  Anxiety will be measured using the Generalized Anxiety Disorder Scale (GAD-7). This self-administered questionnaire consists of seven items, each scored from 0 (not at all) to 3 (nearly every day), with a total score ranging from 0 to 21. Higher scores indicate greater levels of anxiety.
Depression | 20 minutes
  Depression will be assessed using the Patient Health Questionnaire-9 (PHQ-9). This self-administered questionnaire includes nine items, each scored from 0 (not at all) to 3 (nearly every day), with a total score ranging from 0 to 27. Higher scores indicate more severe depression.
Sleep Quality | 20 minutes
  Sleep quality will be evaluated using the Pittsburgh Sleep Quality Index (PSQI). This self-rated questionnaire assesses sleep quality and disturbances over a one-month period. It consists of 19 items, generating seven component scores that are summed to produce a global score ranging from 0 to 21, with higher scores indicating worse sleep quality.
Psychological Well-being | 20 minutes
  Psychological well-being will be assessed using the General Health Questionnaire-12 (GHQ-12). This self-administered questionnaire includes 12 items, each scored on a 4-point scale (less than usual, no more than usual, rather more than usual, or much more than usual), with a total score ranging from 0 to 36. Higher scores indicate greater levels of psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Crisan, PhD, Principal Investigator — University of Medicine and Pharmacy "Victor Babes" Timisoara
Locations (1):
- Spitalul de Boli Infectioase si Pneumoftiziologie Victor Babes, Timișoara, Timiș County, Romania